CLINICAL TRIAL: NCT05130684
Title: Neoadjuvant Nivolumab Plus Paclitaxel/ Cisplatin- Chemo- Radiotherapy (Neo-NTP-CRT) Followed by Esophagectomy for Locally Advanced Esophageal Squamous Cell Carcinoma (ESCC)
Brief Title: Neo-NTP-CRT for Locally Advanced ESCC
Acronym: Neo-NTP-CRT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202005115MIPB
Record Dates: First submitted 2021-10-24; First posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-04

CONDITIONS: Locally Advanced Esophageal Squamous Cell Carcinoma
MeSH Terms: interventions — Nivolumab; Paclitaxel; Cisplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neo-CRT (Experimental): * Nivolumab 240 mg, 30-min IVF, Q2W on days -14, 1, 15, and 29;
  * Paclitaxel 50 mg/m2, 1h-IVF, on days 1, 8, 15, 22, and 29;
  * Cisplatin 30 mg/m2,1h-IVF,on days 1, 8,15, 22, and 29;
  * RT: 1.8 Gy/fraction, 5 days a week, for 25 fractions (total dose= 45 Gy).
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — adding nivolumab to conventional neoadjuvant CRT
  Other Names: paclitaxel; cisplatin; radiation

SUMMARY:
The investigators hypothesize that nivolumab combined with neoadjuvant chemoradiotherapy (CRT) is safe and effective in patients with locally advanced esophageal squamous cell carcinoma (LAESCC).

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven squamous cell carcinoma of the intrathoracic esophagus.
2. Locally advanced disease, which is defined by the TNM system of the American Joint Committee on Cancer (AJCC) Cancer Staging System (8th edition), fulfilling one of the following criteria as determined by endoscopic ultrasound, computed tomography, bronchoscopy and positron emission tomography:

   1. cT3/4a, N0, M0;
   2. cT1-3, N1-3, M0.
3. Tumor length longitudinal ≤ 8cm and radial ≤ 5cm.
4. The tumor must not extend more than 2cm into the stomach.
5. No invasion of the tracheobronchial tree or presence of tracheoesophageal fistula.
6. Age ≥ 20 and ≤ 75 years old.
7. Performance status ECOG 0~1.
8. Adequate bone marrow reserves, defined as:

   1. white blood cells (WBC) ≥ 4,000/µl or neutrophil count (ANC) ≥ 2,000/µl;
   2. platelets ≥ 100,000/µl.
9. Adequate liver function reserves, defined as:

   1. hepatic transaminases ≤ 2.5 x upper limit of normal (ULN);
   2. serum total bilirubin ≤ 2.0 x upper limit of normal (ULN).
10. Adequate renal function: Creatinine ≤1.5 x upper normal limit or estimated creatinine clearance ≥ 50 ml/min (estimated by Cockcroft-Gault formulation)
11. Written informed consent.
12. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
13. Female subjects of childbearing potential must be willing to use an adequate method of contraception as outlined in Section - Contraception, for the course of the study through 120 days after the last dose of study medication.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
14. Male subjects of childbearing potential must agree to use an adequate method of contraception as outlined in Section - Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Adenocarcinoma.
2. Previous thoracic irradiation.
3. Previous systemic chemotherapy
4. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
5. Synchronously diagnosed squamous cell carcinoma of aerodigestive way, other than esophageal cancer.
6. Prior malignancy, except for the following:

   1. adequately treated basal cell or squamous cell skin cancer;
   2. in-situ cervical cancer;
   3. a "cured" malignancy more than 5 years prior to enrollment.
7. Significant co-morbid disease, which prohibits the conduction of chemotherapy, concurrent chemo- radiotherapy, or radical surgery, such as active systemic infection, symptomatic cardiac or pulmonary disease, or psychiatric disorders.
8. Documented myocardial infarction within the 6 months preceding registration (pretreatment ECG evidence of infarct only will not exclude patients). Patients with a history of significant ventricular arrhythmia requiring medication. Patients with a history of 2nd or 3rd degree heart block.
9. Pre-existing motor or sensory neurotoxicity greater than grade 1.
10. Patients with prior allergic reactions to drug containing Cremophor, such as teniposide or cyclosporine.
11. Weight loss > 15%.
12. Dementia or altered mental status that would prohibit the understanding and completion of informed consent.
13. Estimated life expectancy less than 3 months.
14. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
15. Has a known history of active TB (Bacillus Tuberculosis)
16. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
17. Has known history of, or any evidence of active, non-infectious pneumonitis, interstitial lung disease or pulmonary fibrosis.
18. Concurrent diverticulitis or symptomatic gastrointestinal ulcerative disease.
19. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
20. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
21. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., anti-HCV reactive and HCV RNA [qualitative] are detected).
22. Patients with a negative HBs antigen test but a positive test result for either HBs antibody or HBc antibody with a detectable level of HBV-DNA.
23. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
24. Has received organ transplantation.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
change in treatment related death | 30 days
  no increase of treatment-related death within 30 days after esophagectomy
rate of completion of protocol treatment | 5 months
  successful completion of preoperative therapy and processing to surgery without any extended treatment-related delay, which is defined as > 19 weeks after the first dose of nivolumab (d-14) in neo-NTP-CRT (19 weeks include 15 weeks of protocol treatment plus 4 weeks of flexibility.).

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hung Hsu, MD PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No